CLINICAL TRIAL: NCT04157140
Title: Anlotinib Hydrochloride In Combination With Radiofrequency Ablation And Transcatheter Arterial Chemoembolization in Patients With Middle-advanced Hepatocellular Carcinoma, Open, Single Arm, Exploratory Clinical Trial
Brief Title: Anlotinib In Combination With RFA And TACE in Patients With Middle-advanced HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinglong Chen (Other)
Responsible Party: Sponsor-Investigator, Jinglong Chen, Chief of Oncology, Beijing Ditan Hospital
Organization: Beijing Ditan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 320.6750.19089-49
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: anlotinib; HCC; TACE; RFA
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib+ TACE+ RFA (Experimental): Anlotinib+ TACE+ RFA
  Interventions: Drug: Anlotinib; Device: TACE+RFA

INTERVENTIONS:
Drug: Anlotinib — 12mg, continuous oral 2 weeks stop for 1 week, 21 days for a treatment cycle.
Device: TACE+RFA — TACE first, followed by RFA within day7（+/-3days）

SUMMARY:
A single-arm, open-label clinical trial, focus on the safety and efficacy of anlotinib hydrochloride in combination with radiofrequency ablation (RFA) and transcatheter arterial chemoembolization(TACE) in patients with middle-advanced hepatocellular carcinoma(HCC)

ELIGIBILITY:
Inclusion Criteria:

* Patients participate in the study voluntarily and sign informed consent with good compliance.
* Histological or cytological confirmation of unrespectable middle-advanced hepatocellular carcinoma, Barcelona Clinic Liver Cancer stage Category C or B , liver function child-Pugh class A or B (≤7 points).
* At least one measurable lesion, with diameter ≥ 10mm measured by spiral MRI/CT scan per mRECIST; have not received local therapies including but not limited to TACE, RFA, radiotherapy and cryosurgery.-Eastern Cooperative Oncology Group Performance Status 0 or 1.
* Life expectancy of at least 3 months.
* Main organs function is normal. (normal main organs function as defined below: Hemoglobin (Hb) ≥ 90 g/L, Neutrophils (ANC) ≥ 1.5×109/L, leucocyte (WBC) ≥ 3.0×109/L, Platelet count (PLT) ≥ 70×109/L, Total bilirubin (TBIL) ≤ 1.5 × normal upper limit (ULN), Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 ×ULN, Serum creatinine (Cr) ≤ 1.5× ULN or Creatinine Clearance rate(CCr) ≥60ml/min,Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) > 50%)
* The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 3 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 8 weeks after it.
* Patients have disease that is not amenable to potentially curative transplantation or ablation
* Patients who have characterization for targeted therapy treatment, but under poor economic conditions and cannot afford angiogenesis inhibitors recommended by current guidelines, including Lenvatinib, sorafenib, Cabozantinib, Ramolumab, regorafenib, etc.

Exclusion Criteria:

* History of other malignancy within 5 years or for now (except for non-melanoma skin cancer, cervix in situ carcinoma, superficial Bladder neoplasms).
* Subject has obstacle in the function of major organs such as heart, lung, liver and kidney
* Patients who plan liver transplantation.
* Patients who had previously received treatment with target inhibitors or other immunotherapy against or chemotherapy
* Patients who had previously received treatment with TACE or or other local therapy or radiotherapy or Chinese medicine treatment within 4 weeks.
* Liver function status Child-Pugh Class C, with malignant ascites.
* Participated in other anti-tumor clinical trials within 4 weeks.
* Symptoms that affect oral medication and cannot be controlled through proper treatment (such as inability to swallow, chronic diarrhoea and intestinal obstruction, etc.).
* Any of the following coagulation functions are abnormal, including: Prothrombin time (PT)>ULN+4s, Activated partial thromboplastin time (APTT) >1.5ULN s, nternational normalized ratio (INR)>1.5
* Patients who underwent major surgery within 4 weeks.
* Patients who have got non remissive toxic reactions derived from any treatment, which is over level 1 in CTC AE (4.0).
* Patients with any severe and/or unable to control diseases，including： Patients with unsatisfactory blood pressure control using antihypertensive drugs (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100) mmHg); Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QTc≥480ms) and patients with Grade 2 or higher congestive heart failure (NYHA Classification); Patients with active or unable to control serious infections, which is over level 2 in CTC AE (4.0); Patients with poorly controlled diabetes (fasting blood glucose(FBG)>10mmol/L); Patients with kidney failure who require hemodialysis or peritoneal dialysis; Patients with a history of immunodeficiency, including a positive HIV test or other acquired, congenital immunodeficiency disease, or a history of organ transplantation; Urine routine indicates that urine protein ≥ ++, and confirmed 24-hour urine protein quantitation > 1.0 g.
* Patients whose tumors had invaded important blood vessels by imaging or who, as determined by the researchers, were likely to invade important blood vessels during follow-up trial, resulting in fatal bleeding.
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism.
* Regardless of the severity, patients with any physical signs or history of bleeding, patients with bleeding or bleeding events greater than or equal to CTCAE 3 within four weeks prior to the first administration, or patients with unhealed wounds, fractures, ulcers.
* Patients with Brain metastases.
* Patients with cancer thrombus involving whole the main portal vein.
* Female patients who are pregnant or breastfeeding.
* Patients with drug abuse history and unable to get rid of or patients with mental disorders.
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment.
* History of gastrointestinal bleeding due to severe gastroesophageal varices within 4 weeks.
* Severe active or uncontrolled infections.
* Patients who had serious adverse effect to Anlotinib.
* Patients who had serious adverse effect to iodinated contrast agent.
* Liver cirrhosis, hepatic decompensation, active hepatitis or chronic hepatitis which requires anti-viral treatment. Hepatitis C virus (HCV) antibody test shows positive and titer test shows amount of HCV exceeds upper limit of normal (ULN) after treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Time To Progression(TTP) | each 42 days up to progressive disease (PD) (up to 24 months)
  Time To Progression is defined as the time from first day of TACE treatment until the first date of either objective disease progression

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective response rate is defined as the percentage of subjects whose best response was complete response (CR) or partial response (PR) according to the Modified Response Evaluation Criteria in Solid Tumors Version (mRECIST).
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease control rate is defined as the percentage of subjects whose best response was CR, PR or stable disease (SD) according to the mRECIST.
Duration of Response (DOR) | Time Frame: each 42 days up to intolerance the PD or death (up to 24 months)
  Duration of Response is defined as the percentage of subjects whose best response was CR, PR or stable disease (SD) according to the mRECIST or death due to any cause, whichever occurs first.
Incidence of Treatment-Emergent Adverse Events | Until 30 day safety follow-up visit
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - Shengjing Hospital Of China Medical University, Shenyang

IPD SHARING:
Plan to Share IPD: No